CLINICAL TRIAL: NCT01585337
Title: Joint Coordination Changes During Functional Activities After Lumbar Fusion
Brief Title: Trunk Forward Ability in Patients With Lumbar Fusion
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201109033RC
Record Dates: First submitted 2012-04-23; First posted 2012-04-25 (Estimated); Last update posted 2015-07-08 (Estimated); Status verified 2015-07

CONDITIONS: Fusion of Spine, Lumbar Region

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- patients with lumbar fusion

SUMMARY:
The hypotheses of this study are as follows:

1. There is no significant muscle activity difference of each muscle in patients between pre and post operation.
2. There is no significant forward reach distance/average velocity difference in patients between pre and post operation.
3. There is no significant standard deviation of center of pressure (COP) along x axis, speed of COP along y axis during the task and COP path during the 3-sec holding phase difference in patients between pre and post operation.
4. There is no significant muscle activity difference between muscles on both sides at post operation.

DETAILED DESCRIPTION:
30 healthy adults and 30 patients is going to undergo lumbar fusion surgery will be recruited in this study. The assessment will be held before surgery, two months, three months and six months after surgery. Visual pain scale and passive range of motion over lumbar, hip, knee, ankle joint of each subjects will be recorded. Then the maximum voluntary contraction at lower extremity will be measured by electromyography. Finally, the subjects will be asked to do forward reach by dominant upper limb/bilateral upper limbs/arm crossed in the front of chest for three times in standing and sitting position after five practices. The motion data will be collected by 3-dimension video and the muscle activity by electromyography.

ELIGIBILITY:
Inclusion Criteria:

1. specific low back pain with MRI finding by the radiologist and the surgeon;
2. patient who is scheduled for MISS in one week.

Exclusion Criteria:

1. scoliosis;
2. neurological disorder;
3. Self-reported impairment in daily activities;
4. leg length deficiency over 2 cm;
5. body mass index over 30.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All subjects will be recruited from Far Eastern Memorial Hospital. The study is approved by the Institutional Medical Research Ethics Committees in both National Taiwan University Hospital and Far Eastern Memorial Hospital. The consent form is as . We will recruit patients aged between 30 to 60 years old.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2012-01; Primary Completion 2016-02 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
EMG | one months post operation

SECONDARY OUTCOMES:
forward reach distance | one month post operation

CONTACTS AND LOCATIONS:
Overall Officials: Wei-Li Hsu, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University, College of Medicine, Taipei, Taiwan